CLINICAL TRIAL: NCT03161899
Title: Evaluation of Nutritional Status in Patients With Thalassemia Major in Assiut University Children Hospital
Brief Title: Evaluation of Nutritional Status in Thalassemia Major Patients in Assiut Children Hospital
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ARAbdelmonem, resident doctor of pediatrics, Assiut University
Other Study IDs: ENST
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Thalassemia Major
Keywords: thalassemia - nutrition -growth
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thalassemia is a blood disorder passed down through families in which the body makes an abnormal form of hemoglobin. There are 2 main types of thalassemia; Alpha & Beta thalassemia. Alpha thalassemia: occurs when a gene or genes related to the alpha globin protein are missing or mutated.

Beta-thalassemia syndromes are a group of hereditary blood disorders characterized by reduced or absent beta globin chain synthesis. Beta-thalassemias can be classified into:

Silent carrier: completely asymptomatic with normal hematological parameters. Beta-thalassaemia minor (beta-thalassaemia trait): usually asymptomatic; diagnosis is made during a work-up for mild anemia.

Beta-thalassaemia intermedia: usually a similar presentation to beta-thalassaemia major; symptoms are usually less pronounced and the course is usually more insidious.

Beta-thalassaemia major : In which there is complete absence of hemoglobin A

DETAILED DESCRIPTION:
In Egypt beta thalassemia-major is the most common type with carrier rate of 5.3 to ≥9%and 1000 new cases born with beta-thalassemia major per 1.5 million live births per year.

Children born with thalassemia major are normal at birth, but develop severe hemolytic anemia during the first year of life. Symptoms are those of anemia (lethargy, poor feeding, pallor…etc.) failure to thrive and organomegaly. Later on they develop signs of extra medullary hematopoiesis .

Optimal nutritional status is important for growth, immune function, bone health and pubertal development . Various reports suggest the incidence of poor growth ranges from 25% to 75% depending on thalassemia syndrome and severity of disease. This marked growth deficits raise a red ﬂag for any pediatrician to evaluate nutritional status of thalassemic patients and detect possible nutritional deficiencies and associated factors.

Etiology of delayed growth and malnutrition reported in thalassemic patient is multifactorial including :

1. Nutritional deprivation with or without feeding difficulties arising from fatigue and breathlessness
2. Increased energy expenditure secondary to hyper metabolism with or without heart failure
3. Gastrointestinal hypoxia which consequently produces anorexia and malabsorption
4. Reduction of biosynthetic activity of liver.
5. Disturbance of the endocrine function
6. Impaired synthetic hepatic function secondary to hemosiderosis and hepatitis.

The main aim of this study is to assess the nutritional status of thalassemic patient attending Assiut university Children hospital and to determine the factors involved.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed to have thalassemia

Exclusion Criteria:

* patient with any underlaying systemic diseases other than B thalassemia major.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all beta thalassemic patients attending the children Hematology Clinic, Children Hospital, Assiut University, during the period of 1st of June 2017 till 31 th of may 2018.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
percentage of malnutrition | 12 month
  prevalence of malnutrition among thalassemic children attending assiut university children hospital

SECONDARY OUTCOMES:
aetiology poor growth | 12 month
  determination of the most common causes responsible for poor growth seen in thalassemic patients
decrease morbidity | 18 month
  decrease morbidity by providing possible strategies for early prevention of the problem of poor growth occurring in patients with thalassemia major

CONTACTS AND LOCATIONS:
Overall Officials: asmaa refaat, MBBCH, Principal Investigator — Assuit , faculty of medicine, egypt
Locations (1):
- Asmaa Refaat Abdelmonem, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soliman AT, El-Matary W, Fattah MM, Nasr IS, El Alaily RK, Thabet MA. The effect of high-calorie diet on nutritional parameters of children with beta-thalassaemia major. Clin Nutr. 2004 Oct;23(5):1153-8. doi: 10.1016/j.clnu.2004.03.001. PMID 15380908
- [Background] Fung EB. Nutritional deficiencies in patients with thalassemia. Ann N Y Acad Sci. 2010 Aug;1202:188-96. doi: 10.1111/j.1749-6632.2010.05578.x. PMID 20712792
- [Background] Galanello R, Origa R. Beta-thalassemia. Orphanet J Rare Dis. 2010 May 21;5:11. doi: 10.1186/1750-1172-5-11. PMID 20492708